CLINICAL TRIAL: NCT04481191
Title: A Phase 3 Randomized, Open-Label, Clinical Trial to Study the Immunogenicity and Safety of Concomitant and Non-Concomitant Administration of V260 and Inactivated Poliomyelitis Vaccine (IPV) in Chinese Healthy Infants
Brief Title: Immunogenicity and Safety of Concomitant and Non-Concomitant Administration of RotaTeq® (V260) and Inactivated Poliomyelitis Vaccine in Healthy Chinese Infants (V260-074)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V260-074; V260-074 (Other: Merck Protocol Number); 2020-003329-49 (EudraCT Number)
Record Dates: First submitted 2020-07-20; First posted 2020-07-22 (Actual); Results first posted 2023-02-17 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Prevention of Rotavirus Gastroenteritis in Infants and Children Caused by Serotypes G1, G2, G3, G4, and G9
MeSH Terms: interventions — RotaTeq; Rotavirus Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Concomitant RotaTeq and IPV (Experimental): Participants will receive RotaTeq (2 mL oral dose) and IPV (0.5 mL intramuscular [IM] injection ) concomitantly at Visit 2 (15 to 21 days after Visit 1 [Day 1]), Visit 4 (30 to 42 days after Visit 2), and Visit 6 (30 to 42 days after Visit 4).
  Interventions: Biological: RotaTeq (V260); Biological: IPV
- Staggered RotaTeq and IPV (Active Comparator): Participants will receive RotaTeq (2 mL oral dose) at Visit 1 (Day 1), Visit 3 (30 to 42 days after Visit 1), and Visit 5 (30 to 42 days after Visit 3); and IPV (0.5 mL IM injection) at Visit 2 (15 to 21 days Visit 1), Visit 4 (30 to 42 days after Visit 2), and Visit 6 (30 to 42 days after Visit 4).
  Interventions: Biological: RotaTeq (V260); Biological: IPV

INTERVENTIONS:
Biological: RotaTeq (V260) — Live, pentavalent rotavirus vaccine administered as a 2 mL-dose oral solution
  Other Names: RotaTeq; V260
Biological: IPV — 0.5 mL dose IPV (Sabin strain based), administered via IM injection

SUMMARY:
This study will evaluate the immunogenicity and safety of concomitant administration of RotaTeq® (V260) and inactivated poliomyelitis vaccine (IPV) in Chinese infants. Its primary objective is to demonstrate that the immunogenicity of IPV in the concomitant-use group is non-inferior to the immunogenicity of IPV in the staggered-use group. The hypothesis to be tested is: The seroconversion percentage at 1 month post dose 3 for poliovirus types 1, 2, and 3 in the concomitant-use group is non-inferior to those of the staggered-use group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese infant 48 days to 63 days of age.
* Infant's legally acceptable representative provides written informed consent for the study.

Exclusion Criteria:

* History of rotavirus disease, congenital gastrointestinal disorders, chronic diarrhea, failure to thrive, or abdominal surgery.
* History of intussusception.
* History of poliomyelitis.
* Clinical evidence of active gastrointestinal illness. Note: Infants with gastroesophageal reflux disease [GERD] may participate in the study if the GERD is well controlled with or without medication.
* Known or suspected impairment of immunological function, including severe combined immunodeficiency disease (SCID).
* Has a fever, with an axillary temperature ≥37.5°C (or equivalent) at the time of vaccination or within 24 hours prior to vaccination. Note: The Visit 1 may be rescheduled after complete resolution of febrile illness.
* Has acute disease.
* Has underlying diseases such as cardiovascular, renal, liver, or blood disease.
* History of known hypersensitivity to any components of rotavirus vaccine and/or IPV.
* Uncontrolled epilepsy, encephalopathy, seizure, or other progressive neurological diseases.
* Known thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injections.
* Resides in a household with an immunocompromised person, including individuals with congenital immunodeficiency (including SCID), human immunodeficiency virus (HIV) infection, leukemia, lymphoma, multiple myeloma, generalized malignance, chronic renal failure, organ or bone marrow transplantation, or with those receiving immunosuppressive chemotherapy including long-term systemic corticosteroids.
* Any condition, which in the opinion of the investigator, may interfere with the evaluation of the study objectives.
* Prior administration of any rotavirus vaccines or poliovirus vaccines.
* Has received inactivated or recombinant vaccines within 14 days prior to Visit 1 or live vaccines within 28 days prior to Visit 1.
* Has received an investigational or non-registered product other than study vaccines or is planning to use such product during the study.
* Has received immunosuppressive therapies including systemic (intramuscular, oral, or intravenous) corticosteroids. Note: Participants using non-systemic corticosteroids (e.g., topical, ophthalmic, and inhaled) are considered eligible for the study.
* Has received a blood transfusion or blood products, including immunoglobulins or is planning to receive such product during the study.
* Has participated in another interventional study prior to Visit 1 or expected to anytime during the study.
* The infant's legally acceptable representative is unlikely to adhere to the study procedures, keep appointments or is planning to permanently relocate from the area prior to the completion of the study or to leave for an extended period when study visits would need to be scheduled.
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is an investigational site or Sponsor staff member directly involved with this study.

Ages: 48 Days to 63 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-05-08 (Actual); Study Completion 2021-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Yangchun Center For Disease Prevention And Control ( Site 0001), Yangchun, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Chen S, Ying Z, Liu Y, Li Y, Yu Y, Huang M, Huang Z, Ou Z, Liao Y, Zhang Y, Liu G, Zhao W, Fu R, Shou Q, Zheng M, Liao X, Tu Y, Stek J, Hartzel J, Li C, Zhang J. A phase 3 randomized, open-label study evaluating the immunogenicity and safety of concomitant and staggered administration of a live, pentavalent rotavirus vaccine and an inactivated poliomyelitis vaccine in healthy infants in China. Hum Vaccin Immunother. 2024 Dec 31;20(1):2324538. doi: 10.1080/21645515.2024.2324538. Epub 2024 Mar 20. PMID 38509699
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at a study center in China.
Groups:
- Concomitant RotaTeq and IPV: Participants received RotaTeq (2 mL oral dose) and IPV (0.5 mL intramuscular [IM] injection ) concomitantly at Visit 2 (15 to 21 days after Visit 1 [Day 1]), Visit 4 (30 to 42 days after Visit 2), and Visit 6 (30 to 42 days after Visit 4).
- Staggered RotaTeq and IPV: Participants received RotaTeq (2 mL oral dose) at Visit 1 (Day 1), Visit 3 (30 to 42 days after Visit 1), and Visit 5 (30 to 42 days after Visit 3); and IPV (0.5 mL IM injection) at Visit 2 (15 to 21 days Visit 1), Visit 4 (30 to 42 days after Visit 2), and Visit 6 (30 to 42 days after Visit 4).
Period: Overall Study
Arm/Group | Concomitant RotaTeq and IPV | Staggered RotaTeq and IPV
Started | 200 | 200
≥1 V260 Vaccination | 189 | 200
Completed | 185 | 190
Not Completed | 15 | 10
Not completed — Withdrawn by parent/guardian | 15 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Concomitant RotaTeq and IPV | Staggered RotaTeq and IPV | Total
Number analyzed (Participants) | 200 | 200 | 400
Age, Continuous [Mean (Standard Deviation); unit: days] | 53.3 (4.8) | 53.3 (4.6) | 53.3 (4.7)
Age, Customized [Count of Participants; unit: Participants]
  Infants and toddlers (48 to 63 days) | 200 | 200 | 400
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 93 | 179
  Male | 114 | 107 | 221
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 200 | 200 | 400
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 200 | 200 | 400
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Neutralizing Antibody Seroconversion to Poliovirus Types 1, 2, and 3 at 1 Month Post Dose 3 of IPV
Description: The immunogenicity of IPV was measured using poliovirus serum neutralizing antibody assay of the National Institutes for Food and Drug Control (NIFDC), Beijing, China. Serum conversion was defined as antibody titer ≥1:8 post-vaccination in baseline seronegative participants or ≥4-fold increase in titer post-vaccination in baseline seropositive participants.
Time Frame: Baseline and 1 month postdose 3 of IPV (Month ~3.5)
Population: Participants who received the 3 scheduled doses of study vaccination, adhered to guidelines for vaccine administration, provided baseline and post-vaccination blood samples within the acceptable day range, and did not have important protocol deviations are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Concomitant RotaTeq and IPV | Staggered RotaTeq and IPV
Number analyzed (Participants) | 180 | 187
Percentage of Participants
  Poliovirus Type 1 | 98.9 | 100.0
  Poliovirus Type 2 | 98.3 | 99.5
  Poliovirus Type 3 | 100.0 | 99.5
Statistical Analysis 1: Comparison: Concomitant RotaTeq and IPV vs Staggered RotaTeq and IPV; Difference indicates Concomitant-use Group % - Staggered-use Group %; Test type: Non-Inferiority — Non-inferiority was declared when the lower bound of the 95% CI for the difference in percentages (Concomitant-use Group - Staggered-use Group) being > -10 percentage points (one-sided p-value < 0.025); p < 0.001, Unstratified Miettinen & Nurminen method — One-sided p-value; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-4.0 to 0.9]
Statistical Analysis 2: Comparison: Concomitant RotaTeq and IPV vs Staggered RotaTeq and IPV; Difference indicates Concomitant-use Group % - Staggered-use Group %; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Unstratified Miettinen & Nurminen method — One-sided p-value; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-4.3 to 1.5]
Statistical Analysis 3: Comparison: Concomitant RotaTeq and IPV vs Staggered RotaTeq and IPV; Difference indicates Concomitant-use % - Staggered-use %; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Unstratified Miettinen & Nurminen method — One-sided p-value; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-1.6 to 3.0]

2. Secondary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibody to Poliovirus Types 1, 2, and 3 at 1 Month Post Dose 3 of IPV
Description: The immune response to IPV was measured using poliovirus serum neutralizing antibody assay of the NIFDC, Beijing, China.
Time Frame: 1 month postdose 3 of IPV (Month ~3.5)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Concomitant RotaTeq and IPV | Staggered RotaTeq and IPV
Number analyzed (Participants) | 180 | 187
Titers
  Poliovirus Type 1 | 5600.80 (4898.46) [4898.46 to 6403.85] | 5344.24 (4657.51) [4657.51 to 6132.22]
  Poliovirus Type 2 | 1059.83 (951.13) [951.13 to 1180.96] | 1122.43 (1002.74) [1002.74 to 1256.41]
  Poliovirus Type 3 | 3405.56 (3033.93) [3033.93 to 3822.71] | 3261.69 (2913.70) [2913.70 to 3651.24]

3. Secondary Outcome: Percentage of Participants Achieving Neutralizing Antibody Titers ≥1:8 for Poliovirus Types 1, 2, and 3 at 1 Month Post Dose 3 of IPV
Description: The immune response to IPV was measured using poliovirus serum neutralizing antibody assay of the NIFDC, Beijing, China.
Time Frame: 1 month post dose 3 of IPV (Month ~3.5)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Concomitant RotaTeq and IPV | Staggered RotaTeq and IPV
Number analyzed (Participants) | 180 | 187
Percentage of Participants
  Poliovirus Type 1 | 100.0 (98.0) [98.0 to 100.0] | 100.0 (98.0) [98.0 to 100.0]
  Poliovirus Type 2 | 100.0 (98.0) [98.0 to 100.0] | 100.0 (98.0) [98.0 to 100.0]
  Poliovirus Type 3 | 100.0 (98.0) [98.0 to 100.0] | 100.0 (98.0) [98.0 to 100.0]

4. Secondary Outcome: Percentage of Participants Achieving Neutralizing Antibody Titers ≥1:64 for Poliovirus Types 1, 2, and 3 at 1 Month Post Dose 3 of IPV
Description: The immune response to IPV was measured using poliovirus serum neutralizing antibody assay of the NIFDC, Beijing, China.
Time Frame: 1 month postdose 3 of IPV (Month ~3.5)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Concomitant RotaTeq and IPV | Staggered RotaTeq and IPV
Number analyzed (Participants) | 180 | 187
Percentage of Participants
  Poliovirus Type 1 | 100.00 (98.0) [98.0 to 100.0] | 100.0 (98.0) [98.0 to 100.0]
  Poliovirus Type 2 | 100.0 (98.0) [98.0 to 100.0] | 100.0 (98.0) [98.0 to 100.0]
  Poliovirus Type 3 | 100.0 (98.0) [98.0 to 100.0] | 100.0 (98.0) [98.0 to 100.0]

5. Secondary Outcome: Percentage of Participants With Solicited Injection-Site Adverse Events
Description: Solicited injection-site adverse events (AEs) included erythema, swelling, induration, and pain at the IPV injection-site.
Time Frame: Up to 7 days following each IPV vaccination
Population: All participants who received ≥1 dose of study treatment are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Concomitant RotaTeq and IPV | Staggered RotaTeq and IPV
Number analyzed (Participants) | 189 | 200
Percentage of Participants | 25.4 | 23.0

6. Secondary Outcome: Percentage of Participants With Solicited Systemic Adverse Events
Description: Solicited systemic AEs included diarrhea, vomiting, and elevated temperature (axillary temperature ≥37.5º C).
Time Frame: Up to 7 days following each RotaTeq and/or IPV vaccination
Population: All participants who received ≥1 dose of study treatment and have data available are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Concomitant RotaTeq and IPV | Staggered RotaTeq and IPV
Number analyzed (Participants) | 189 | 200
Percentage of Participants
  Elevated temperature: number analyzed (Participants) | 187 | 196
  Elevated temperature | 12.3 | 16.3
  Diarrhoea | 13.2 | 21.5
  Vomiting | 10.6 | 19.5

7. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: The percentage of participants with SAEs is presented. An SAE is an AE that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or another important medical event.
Time Frame: Up to approximately 3.5 months
Population: All participants who received ≥1 dose of study treatment are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Concomitant RotaTeq and IPV | Staggered RotaTeq and IPV
Number analyzed (Participants) | 189 | 200
Percentage of Participants | 3.7 | 5.5

ADVERSE EVENTS:
Time Frame: Up to approximately 3.5 months
Description: All participants who received ≥1 study-related vaccination are included.
Arm/Group | Concomitant RotaTeq and IPV | Staggered RotaTeq and IPV
All-Cause Mortality (participants affected / at risk) | 0/189 | 0/200
Serious Adverse Events (participants affected / at risk) | 7/189 | 11/200
Other Adverse Events (participants affected / at risk) | 123/189 | 143/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concomitant RotaTeq and IPV (N=189) | Staggered RotaTeq and IPV (N=200)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 6 (6)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Motor developmental delay (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concomitant RotaTeq and IPV (N=189) | Staggered RotaTeq and IPV (N=200)
Diarrhoea (Gastrointestinal disorders) | 33 (43) | 50 (77)
Dyspepsia (Gastrointestinal disorders) | 10 (13) | 13 (14)
Vomiting (Gastrointestinal disorders) | 20 (23) | 39 (66)
Injection site erythema (General disorders) | 45 (62) | 41 (45)
Injection site pain (General disorders) | 12 (14) | 7 (7)
Pyrexia (General disorders) | 30 (33) | 37 (48)
Bronchitis (Infections and infestations) | 8 (9) | 13 (14)
Upper respiratory tract infection (Infections and infestations) | 31 (40) | 36 (41)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (26) | 14 (16)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 18 (20)
Eczema (Skin and subcutaneous tissue disorders) | 14 (14) | 12 (18)
Nasopharyngitis (Infections and infestations) | 14 (14) | 14 (16)

LIMITATIONS AND CAVEATS:
Protocol Amendment 3 was issued after study completion. The purpose of the amendment was to update the Sponsor entity name and address.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT04481191/Prot_SAP_000.pdf